CLINICAL TRIAL: NCT02511080
Title: Effectiveness of Spot-on ™ to Prevent Inadvertent Perioperative Hypothermia and Their Consecuences
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osakidetza (Other)
Responsible Party: Principal Investigator, Unai Ortega Mera, Doctor, Osakidetza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEIC 16/2015
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2015-08

CONDITIONS: Hypothermia
Keywords: Spot-on; perioperative hypothermia.
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spot-on group (Active Comparator): Use active measures against intraoperative hypothermia
  Interventions: Device: Spot-On
- control (No Intervention): standard measures against intraoperative hipothermia

INTERVENTIONS:
Device: Spot-On — use of active hot measures
  Arms: Spot-on group

SUMMARY:
Using the spot-on device for monitoring core body temperature during colon laparoscopic surgery and prevent non-therapeutic hypothermia.

DETAILED DESCRIPTION:
Take active measures to prevent non-therapeutic hypothermia during the laparoscopic colon surgery. We improve these measures using heat conductive air warm blankets placed under and o over the patient.

Perform monitoring core body temperature every 15 minutes by spot-on device compared with standard nasopharyngeal probe.

ELIGIBILITY:
Inclusion Criteria:

* All patients that need a colorrectal laparoscopic surgery

Exclusion Criteria:

* Use of antagonist of Calcium
* Alergy to medications
* History of Malignant Hipertemia
* Laparosocopy surgery ≥ 120 min
* Temperature previous surgery over 38ºC
* Taking chronic steroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change in the Body Core Temperature | measure every 15 minutes since the patient arrive to operating room until is derivated to recovery room, an average of 3 hours
  measure the body core temperature by Spoton device when the patient arrive to operating room

SECONDARY OUTCOMES:
incidence of blood transfusion | In the first two weeks after being operated.
  Transfusion if hemoglobin lower than 7 mgr/dl
surgical wound infection | while the patient stay in the hospital, an average of two weeks
  the surgeon determines the infection of the surgical wound

CONTACTS AND LOCATIONS:
Overall Officials: unai ortega, Principal Investigator — Osakidetza
Locations (1):
- Hospital de Galdakao, Galdakao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Torossian A. Thermal management during anaesthesia and thermoregulation standards for the prevention of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):659-68. doi: 10.1016/j.bpa.2008.07.006. PMID 19137809
- [Background] Eshraghi Y, Nasr V, Parra-Sanchez I, Van Duren A, Botham M, Santoscoy T, Sessler DI. An evaluation of a zero-heat-flux cutaneous thermometer in cardiac surgical patients. Anesth Analg. 2014 Sep;119(3):543-549. doi: 10.1213/ANE.0000000000000319. PMID 25045862